CLINICAL TRIAL: NCT01172171
Title: Intracoronary Injection of Melatonin for Patients With ST-elevation Myocardial Infarction: a Placebo Controlled Randomized Study
Brief Title: The Effect of Melatonin on Ischemia-reperfusion Injury Following Acute Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Ismail Gögenür, MD, DMSc, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NLH-01
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Acute Myocardial Infarction; Ischemia-reperfusion Injury
Keywords: Ischemia-reperfusion injury; Acute Myocardial Infarction; Intracoronary melatonin
MeSH Terms: conditions — Reperfusion Injury | interventions — Melatonin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Active Comparator): The randomized patients will receive 10 ml 0,1 mg/ml melatonin intracoronarily and 49 mg intravenously.
  Interventions: Drug: Melatonin, N-acetyl-5-methoxytryptamine
- Isotonic saline (Placebo Comparator): The randomized patients will receive 10 ml isotonic saline (NaCl)and 490 ml intravenously.
  Interventions: Drug: Isotonic saline, Natrium chloride

INTERVENTIONS:
Drug: Melatonin, N-acetyl-5-methoxytryptamine — The investigators will give the randomized patients 10 ml of 0,1 mg/ml melatonin intracoronarily and 490 ml of 0,1 mg/ml (49 mg) melatonin.
  Arms: Melatonin
Drug: Isotonic saline, Natrium chloride — The randomized patients will be given 10 ml of isotonic saline intracoronarily and 490 ml intravenously.
  Arms: Isotonic saline

SUMMARY:
In Denmark, 12.000 people a year, is struck by acute myocardial infarction. A third of these cannot be saved before treatment is possible.

Despite quick and effective reperfusion of the coronary arteries using PCI (Percutaneous Coronary Intervention) after an acute ST-elevation myocardial infarction, substantial morbidity and mortality remain. Infarct size is an important determinant of the short-and long-term outcome after acute myocardial infarction. The most widely used and most effective proven therapy to limit infarct size is the early reperfusion induced by or PCI.

Although beneficial in terms of myocardial salvage, reperfusion itself may contribute to additional damage of the myocardium; the damage due to the combined processes is known as "ischemia-reperfusion injury". The pathogenesis of myocardial ischemia-reperfusion injury is a multifactorial process involving the interaction of multiple mechanisms. Numerous studies indicate that there are three pivotal factors in the pathogenesis of ischemia-reperfusion injury: elevated oxidative damage, depressed energy metabolism, and altered calcium homeostasis.

Partially reduced species of oxygen, including the superoxide anion radical, hydroxyl radical, and hydrogen peroxide, are generated intracellularly as by-product of oxygen metabolism. These reactive oxygen species cause peroxidation af membrane lipids, denaturation of proteins, and modification of DNA, all of which ultimately can lead to cell death. In mammals, cell damage induced by partially reduced oxygen species can also initiate local inflammatory responses, which then lead to further oxidant-mediated tissue injury.

Melatonin is mainly known for its role as an endogenously produced circadian hormone.

For the last twenty years, increasing evidence has proven melatonin to be a very potent direct and indirect antioxidant.

Recent experimental studies have documented the beneficial effects of melatonin in reducing tissue damage and limiting cardiac pathophysiology in models of experimental ischemia-reperfusion.

Primary hypothesis: Melatonin given to patients undergoing PCI can reduce the myocardial damage sustained by ischemia-reperfusion.

DETAILED DESCRIPTION:
Purpose The purpose of this Ph.D study is to examine the antioxidative effect of melatonin in relation to ischemia-reperfusion injury.

The investigators wish to examine to which extend melatonin administered to patients undergoing primary PCI for acute myocardial infarction will reduce the damage of the myocardium caused by ischemia-reperfusion injury and thereby hopefully improve the clinical outcome.

Theory and hypotheses Because there is strong evidence that free radicals contribute to post-ischemic injury, antioxidant enzyme therapy could potentially be extremely effective in reducing the cellular damage. In reality, however, the usefulness of this therapy is limited by a number of factors, in particular the ability of the antioxidants to penetrate the cell membrane and to scavenge free radicals in situ. Fortunately, this limitation can, in part, be addressed with the use of melatonin, a potent indirect and direct free radical scavenger that easily diffuses through the cell membrane to exert its antioxidant effects in all compartments of the cell. Indeed, in contrast to the partial of distribution of other antioxidants, such as vitamin C or E, the melatonin distributes it readily in all subcellular compartments owing to its double-solubility in both, aqueous and in lipid environment. Several recent publications present evidence that the newly discovered antioxidant melatonin has significant protective actions against the cardiac damage such as occurs during ischemia-reperfusion injury.

Primary hypothesis: Melatonin given to patients undergoing PCI can reduce the myocardial damage sustained by ischemia-reperfusion.

Inclusion:

* Adults who are able to give informed consent
* 1 significant coronary occlusion (>2mm) with TIMI 0-1 expected to undergo PCI.
* ECG criteria: The occlusion must be ECG-verified with new ST-elevations ≥ 0.2 mV in V2-V3 and/or ≥ 0.1 in the other leads or with a new onset left bundle branch block.
* Having onset of symptoms of qualifying AMI and undergo PCI within 6 hours.
* If the patients do not fulfill the ECG inclusion criteria they can still be included if the primary PCI reveals an acute coronary occlusion (>2mm) with TIMI 0-1.

Exclusion: Patients with prior myocardial infarction, more than one significant occlusion, prehospital thrombolysis, known history of renal failure, history of autoimmune diseases, pregnancy, fertile women or breastfeeding, severe concurrent illness with reduced short-term prognosis, pacemaker, claustrophobia, cardiogenic shock, metals in the body, atrial fibrillation, BMI ≥ 40.

Intervention: The STEMI patient with 1 significant occlusion undergoing PCI less than 6 hours from onset of symptoms will be randomized to intracoronary injection of either melatonin or placebo(saline). The melatonin or placebo will be given as a bolus of 10 ml in relation to PCI, as soon as the occlusion is removed. Immediately after the bolus is given, a solution of 490 ml of either placebo (saline) or 0,1 mg/ml melatonin (49 mg melatonin)will be given intravenously over 6 hours (80 ml/hour).

Primary end point: MRI of the heart at day 4 (+/- 1 day) after the PCI procedure to determine myocardial salvage index.

Secondary end point:

* To determine whether melatonin treatment reduces infarct size as determined by the concentration of high sensitive TnT or high-sensitive TnI and Creatinin Kinase Myocardial Band (CK-MB)(area under the curve) in the blood, measured daily for the first 4 days after AMI.
* the concentration of plasma melatonin after PCI
* the concentration of oxidative markers 24 hours after PCI

Clinical events occurring within the first 90 days after surgery; death, sustained ventricular arrhythmias, resuscitation from cardiac arrest, cardiogenic shock, heart failure, major bleedings, stroke, need for revascularization, recurrent ischemia, re-infarctions and re-hospitalization.

Design: Randomized, double-blind, placebo-controlled interventional study.

Method: Patients who meet the criteria of inclusion will be randomized to intra-coronary injection plus intravenous infusion of melatonin or placebo. The bolus will be given just after the opening of the vessel (TIMI ≥ 2) . Hs-Troponin T/I and CK-MB will be measured in a blood sample taken 1 hour, 6 hours, 24 hours, 48 hours, 72 hours and 96 hours after the PCI procedure. At day 4 after PCI, the patients will undergo MRI of the heart focusing on infarct size and area at risk.

Patient number: Statistical power analysis shows that with a type 1 error of 5% and a type 2 error of 20%, mean at 9,63 and the SD with MRI of 0,16, one should be able to detect a difference in infarct size of 25% between the two groups, when including 2x17 patients in each group. The investigators are including 2x 20 patients.

Safety: The experiments are considered to be of no risk or discomfort for the patients. Both the intervention group and the placebo group are operated by current clinical guidelines.

ELIGIBILITY:
Inclusion criteria:

* Adults who are able to give informed consent
* 1 significant coronary occlusion (>2mm) with TIMI 0-1 expected to undergo PCI.
* The occlusion must be ECG-verified with new ST-elevations ≥ 0.2 mV in V2-V3 and/or ≥ 0.1 in the other leads or a new onset left bundle branch block.
* Having onset of symptoms of qualifying AMI and undergo PCI within 6 hours.
* If the patients do not fulfill the ECG inclusion criteria they can still be included if the primary PCI reveals an acute coronary occlusion (>2mm) with TIMI 0-1.

Exclusion criteria:

* Patients with prior myocardial infarction
* more than one significant occlusion
* prehospital thrombolysis
* known history of renal failure
* history of autoimmune diseases
* pregnancy, fertile women or breastfeeding
* severe concurrent illness with reduced short-term prognosis
* pacemaker
* claustrophobia
* cardiogenic shock
* metals in the body
* atrial fibrillation
* BMI ≥ 40.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
MRI of the heart | day 4 after pci (+/- 1 day)
  Focusing on quantification infarct size, area at risk and myocardial salvage index

SECONDARY OUTCOMES:
Creatinin Kinase Myocardial Band (CK-MB) | 96 Hours after pci
  CK-MB is a cardiac enzyme, which is elevated when the myocardium is damaged.
Clinical events | Within 90 days of pci
  Death, sustained ventricular arrhythmias, resuscitation from cardiac arrest, cardiogenic shock, heart failure, major bleedings, stroke, need for revascularization, recurrent ischemia, re-infarctions and re-hospitalization.
High-sensitive Troponin T (Hs-TnT) or High-sensitive TnI | 96 hours after pci
  Troponin T/I is a cardiac enzyme, which rises when the myocardium is damaged. To determine whether melatonin treatment reduces infarct size as determined by the concentration of Troponin T/I (area under the curve) in the blood, it will be measured daily for the first 4 days after infarction.
plasma level of melatonin | after pci
  An assessment of the endogenous level of plasma melatonin
Oxidative markers in plasma | 24 hours after pci

CONTACTS AND LOCATIONS:
Overall Officials: Ismail L. Gögenur, MD, DSMc, Principal Investigator — Herlev Hospital
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg, Aalborg
  - Odense University Hospital, Odense, Odense

REFERENCES:
- [Derived] Halladin NL, Busch SE, Jensen SE, Hansen HS, Zaremba T, Aaroe J, Rosenberg J, Gogenur I. Intracoronary and systemic melatonin to patients with acute myocardial infarction: protocol for the IMPACT trial. Dan Med J. 2014 Feb;61(2):A4773. PMID 24495883